CLINICAL TRIAL: NCT02332954
Title: Interventional, Open-Label, Single Cohort, Canadian Study to Describe the Relationship Between Cognitive Symptoms and Work Productivity in Working Adults Treated With Vortioxetine for Major Depressive Disorder (MDD)
Brief Title: Assessment in Work Productivity and the Relationship With Cognitive Symptoms in Patients With MDD Taking Vortioxetine
Acronym: AtWoRC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundbeck Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15913A
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Cognition; Cognitive symptoms; vortioxetine; real life; naturalistic
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Neurobehavioral Manifestations | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vortioxetine naive (Other): vortioxetine 10 mg 100 patients with Major Depressive Disorder who have not been treated with another antidepressant for the current MDE
  Interventions: Drug: vortioxetine
- Switch (Other): vortioxetine 10 mg 100 patients with Major Depressive Disorder that require a switch from their current antidepressant due to inadequate response
  Interventions: Drug: vortioxetine

INTERVENTIONS:
Drug: vortioxetine — The starting and recommended dose of vortioxetine is 10 mg once daily; film-coated 10 mg tablets for oral use once daily for 52 weeks.Depending on individual patient response, the dose may be increased to a maximum of 20 mg daily.
  Other Names: Trintellix

SUMMARY:
The purpose of the study is to describe the association/correlation between change in patient-reported cognitive symptoms and work productivity in gainfully employed patients receiving vortioxetine for a Major Depressive Episode (MDE).

DETAILED DESCRIPTION:
This is an interventional, Canadian, multi-site, open-label, single cohort, flexible-dose study. The study will emulate a naturalistic real-life setting. Investigators will include Primary Care Physicians and Psychiatrists working in outpatient clinics. The study will include adult patients diagnosed with MDD according to the DSM-5™. Approximately 200 patients will be enrolled in the study. There will be approximately 100 patients who receive vortioxetine as a first treatment for the current MDE and 100 patients switched to vortioxetine due to inadequate response to their current antidepressant medication treatment. All patients will be treated with vortioxetine as per the product monograph, and at the doses determined appropriate by the investigator. The total study duration from Baseline to the end of follow-up will be approximately 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a man or woman, aged ≥18 years and <65 years (In the province of British Columbia, the patient must be aged 19 years or older in order to give Informed Consent)
* The patient is engaged in volunteer work or gainful employment (working ≥20 hours per week) or is enrolled full-time in post-secondary studies or vocational training.
* The patient is an outpatient consulting a Primary Care Physician or a Psychiatrist.
* Patients must have a diagnosis of MDD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5™) classification code 296.3x.
* The current MDE is confirmed by the investigator.
* The reported duration of the current MDE is at least 3 months.
* The patient has a Baseline score ≥15 on the QIDS-SR.
* The patient reports at least a minimal level of cognitive symptoms as defined by Baseline score of ≥30 on the PDQ-D-20.
* The patient is capable of communicating with the site personnel and is able to conduct the digit-symbol substitution test (DSST).

Exclusion Criteria:

* The patient score is >69 on the DSST at Screening/Baseline.
* The patient is, in the opinion of the investigator, not able to complete all the study assessments including, but not limited to, patient-reported assessments and the DSST.
* The patient has a current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features.
* The current depressive symptoms are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each at the maximum recommended dose (according to Canadian labeling).

Other protocol defined inclusion and exclusion criteria do apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-02; Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
the association/correlation between changes in patient-reported cognitive symptoms and work productivity. (Perceived Deficit Questionnaire-Depression) | 12 weeks
  Mean change from Baseline to Week 12 in patient-reported cognitive symptoms as measured by Perceived Deficit Questionnaire-Depression-20 questions (PDQ-D-20) and work productivity as measured by Work Limitations Questionnaire (WLQ) in gainfully employed patients receiving vortioxetine for a Major Depressive Episode (MDE).

SECONDARY OUTCOMES:
Cognitive function (PDQ-D-20) | 12 and 52 weeks
  Mean change from baseline in cognitive symptoms as measured by PDQ-D-20.
Cognitive function (Digit Symbol Substitution Test (DSST) | 12 and 52 weeks
  Mean change from baseline in cognitive symptoms as measured by Digit Symbol Substitution Test (DSST).
Work productivity (WLQ) | 12 and 52 weeks
  mean change from baseline in work productivity as measured by WLQ.
Work productivity (Work Productivity and Activity Impairment (WPAI) questionnaire) | 12 and 52 weeks
  mean change from baseline in work productivity as measured by Work Productivity and Activity Impairment (WPAI) questionnaire.
Work productivity (World Health Organization Disability Assessment Schedule-12 questions (WHODAS-12) | 12 and 52 weeks
  mean change from baseline in work productivity as measured by World Health Organization Disability Assessment Schedule-12 questions (WHODAS-12).
Work productivity (Sheehan Disability Scale (SDS) | 12 and 52 weeks
  mean change from baseline in work productivity as measured by Sheehan Disability Scale (SDS).
Depressive symptoms (Quick Inventory of Depression Symptomatology-Self Report (QIDS-SR) | 12 and 52 weeks
  mean change from baseline in depressive symptoms as measured by Quick Inventory of Depression Symptomatology-Self Report (QIDS-SR).
Depressive symptoms (Clinical Global Impression-Improvement (CGI-I) score) | 12 and 52 weeks
  mean change in depressive symptoms as measured by Clinical Global Impression-Improvement (CGI-I) score.
Depressive symptoms (Clinical Global Impression-Severity (CGI-S) | 12 and 52 weeks
  mean change from baseline in depressive symptoms as measured by Clinical Global Impression-Severity (CGI-S).

CONTACTS AND LOCATIONS:
Overall Officials: Pratap Chokka, M.D., Principal Investigator — Chokka Center for Integrative Health
Locations (26):
- Canada (26):
  - CA004, Edmonton, Alberta
  - CA005, Kelowna, British Columbia
  - CA006, St. John's, Newfoundland and Labrador
  - CA007, Halifax, Nova Scotia
  - CA016, Burlington, Ontario
  - CA013, Chatham, Ontario
  - CA010, Corunna, Ontario
  - CA012, Fort Erie, Ontario
  - CA017, Hamilton, Ontario
  - CA026, Hamilton, Ontario
  - CA011, London, Ontario
  - CA003, Mississauga, Ontario
  - CA008, Sarnia, Ontario
  - CA009, Sarnia, Ontario
  - CA015, St. Catharines, Ontario
  - CA022, Montreal, Quebec
  - CA020, Montreal, Quebec
  - CA023, Montreal, Quebec
  - CA018, Pointe-Claire, Quebec
  - CA024, Saint-Jean-sur-Richelieu, Quebec
  - CA030, Victoriaville, Quebec
  - CA027, Westmount, Quebec
  - CA028, Saskatoon, Saskatchewan
  - CA019, Québec
  - CA021, Québec
  - CA029, Québec

REFERENCES:
- [Derived] Chokka P, Bougie J, Proulx J, Tvistholm AH, Ettrup A. Long-term functioning outcomes are predicted by cognitive symptoms in working patients with major depressive disorder treated with vortioxetine: results from the AtWoRC study. CNS Spectr. 2019 Dec;24(6):616-627. doi: 10.1017/S1092852919000786. PMID 30802419